CLINICAL TRIAL: NCT01860924
Title: Supervised, Vigorous Intensity Exercise Intervention for Depressed Female Smokers
Brief Title: Vigorous Exercise for Depressed Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christi Patten, Professor of Psychology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-006106
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Nicotine Dependence; Depression
Keywords: exercise; depression; smoking
MeSH Terms: conditions — Tobacco Use Disorder; Depression; Motor Activity; Smoking | interventions — Exercise; Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- health education (Active Comparator): health education control
  Interventions: Behavioral: health education
- exercise (Experimental): vigorous supervised exercise
  Interventions: Behavioral: exercise

INTERVENTIONS:
Behavioral: exercise — vigorous intensity exercise
  Other Names: physical activity
  Arms: exercise
Behavioral: health education — education
  Other Names: health
  Arms: health education

SUMMARY:
In this project the investigators will develop and pilot test a supervised, vigorous intensity exercise intervention for depressed female smokers. If the pilot intervention is successful the investigators will have a blueprint for a large randomized controlled trial. The long term objective is to develop interventions for depressed women that will ultimately reduce their risk of tobacco-caused disease and mortality.

DETAILED DESCRIPTION:
This project will be the first to evaluate supervised vigorous exercise for depressed smokers

ELIGIBILITY:
INclusion Criteria:

1. depressed (CES-D) score 16 or above
2. 18 years of age
3. female gender
4. sedentary
5. current cigarette smoker

Exclusion Criteria:

1. smoking cessation medication
2. Not able to exercise medically

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
smoking abstinence | 6 months
  Smoking cessation biochemically confirmed

SECONDARY OUTCOMES:
depressive symptoms | 6 months
  depressive symptoms (PHQ-9)

CONTACTS AND LOCATIONS:
Overall Officials: Christi Patten, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902